CLINICAL TRIAL: NCT05571865
Title: Preventing Diabetic Cardiomyopathy and Heart Failure by Ketone Bodies
Brief Title: Diabetic Cardiomyopathy and Heart Failure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not receive funding as anticipated.
Sponsor: University of Louisville (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00002; PA-20-190 (Other: NIH)
Record Dates: First submitted 2022-09-16; First posted 2022-10-07 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Diabetic Cardiomyopathies; Heart Failure
Keywords: Diabetic Cardiomyopathy, Metabolic Dysregulation, and Heart Failure.
MeSH Terms: conditions — Diabetic Cardiomyopathies; Heart Failure | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Diabetic, and non-diabetic subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control subjects (non-diabetic). (Other): Control subjects (non-diabetic):
  10 subjects: No intervention (placebo). 10 subjects: Intervention (probiotic)
  Interventions: Dietary Supplement: Probiotic
- Diabetic Subjects (Other): Diabetic subjects:
  10 subjects: No intervention (placebo). 10 subjects: Intervention (probiotic)
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — Oral administration of a probiotic

SUMMARY:
This study will demonstrate the beneficial effects of ketone bodies in type 1 diabetes (T1D) patients and will have significant translational applications to prevent serious metabolic conditions such as T1D induced diabetic cardiomyopathy (DCM).

DETAILED DESCRIPTION:
T1D remains the primary cause of DCM. The long-term goal is to understand the mechanism of T1D leading to DCM. Proprotein convertase subtilisin/kexin type 9 (PCSK9) plays an important role in degrading the low-density lipoprotein receptors (LDLRs) and that increases the circulating LDL cholesterol (LDL-C). Further, PCSK9 increases duringT1D and that, in turn, decreases mitochondrial bioenergetics, transcription factor- mitochondrial (TFAM), and the mitochondrial numbers thus creates an oxidative stress. These changes lead to oxidation of high-density lipoprotein paraoxonase-1 (HDL-Pon1). Because Pon1 hydrolyzes homocysteine (Hcy), the oxidized Pon1 thus causes accumulation of Hcy (i.e. hyperhomocysteinemia; HHcy). Also, the 'metabolic memory' is associated with epigenetic modification (methylation) of genes encoding proteins such as thioredoxin interacting protein (TXNIP). Since methylation/epigenetics inhibits genes, this phenomenon generates even more amounts of Hcy. Investigators have shown that HHcy decreases G-protein coupled receptor (GPCR) Gαs subunit, protein kinase-B (AKT), focal adhesion kinase (FAK) but increases calpain-1, inflammasome and oxidative stress. The central hypothesis is that an increase in PCSK9 causes oxidative stress and decreases TXNIP thus causing oxidation of HDL-Pon1 and subsequent accumulation of Hcy. These alterations lead to decrease in Gαs, AKT, FAK and concomitant increase in PCSK9 and calpain-1 causing metabolic, diastolic, and systolic cardiac dysfunction. Treatment with ketone bodies (the food for mitochondria) will mitigate these changes.

ELIGIBILITY:
Inclusion Criteria:

-Diabetic subjects with high blood glucose levels

Exclusion Criteria:

- Comorbidities affecting glucose levels and cardiac function

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Both male and female representing race/ethnicity
Enrollment: 0 (Actual)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure-I | 4 years
  Levels of glucose in blood and urine
Primary Outcome Measure-II | 4 years
  Cardiac function evaluation by electrocardiogram

SECONDARY OUTCOMES:
Secondary Outcome Measure-I | 4 years
  Biochemical estimation of biomarkers from blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Mahavir Singh, DVM, MS, PhD, Principal Investigator — University of Louisville School of Medicine
Locations (1):
- University of Louisville School of Medicine, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
Outcomes of the probiotic intervention in diabetic patients for the prevention of cardiomyopathy.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: As soon as the data is collected, and fully analyzed.
Access Criteria: Via personal meetings, national and international conferences.

REFERENCES:
- [Result] Mishra SP, Wang S, Nagpal R, Miller B, Singh R, Taraphder S, Yadav H. Probiotics and Prebiotics for the Amelioration of Type 1 Diabetes: Present and Future Perspectives. Microorganisms. 2019 Mar 2;7(3):67. doi: 10.3390/microorganisms7030067. PMID 30832381
- [Result] Wang CH, Yen HR, Lu WL, Ho HH, Lin WY, Kuo YW, Huang YY, Tsai SY, Lin HC. Adjuvant Probiotics of Lactobacillus salivarius subsp. salicinius AP-32, L. johnsonii MH-68, and Bifidobacterium animalis subsp. lactis CP-9 Attenuate Glycemic Levels and Inflammatory Cytokines in Patients With Type 1 Diabetes Mellitus. Front Endocrinol (Lausanne). 2022 Mar 1;13:754401. doi: 10.3389/fendo.2022.754401. eCollection 2022. PMID 35299968